CLINICAL TRIAL: NCT01949558
Title: From Efficacy to Effectiveness: Randomized Controlled Trial of Lifestyle Intervention Postpartum Among Overweight and Obese Women Within Primary Health Care in the Vastra Gotaland Region
Brief Title: Randomized Controlled Trial of Lifestyle Intervention Postpartum in Primary Health Care
Acronym: LIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIV 2011-0193; FORTE LIV (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2013-09-20; First posted 2013-09-24 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Overweight; Obesity
Keywords: diet; lifestyle
MeSH Terms: conditions — Overweight; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group receives a brochure on healthy dietary habits according to regular care.
- Dietary intervention (Experimental): 12 week individual intervention based on a cognitive behavioral approach. It includes dietary restriction under guidance by a dietitian. Thereafter monthly follow-up takes place via email during the following 9 mo.
  Interventions: Behavioral: Dietary Intervention

INTERVENTIONS:
Behavioral: Dietary Intervention
  Arms: Dietary intervention

SUMMARY:
Chronic diseases such as overweight and cardiovascular diseases represent important threats to women's health. Pregnancy and lactation are associated with changes in weight, body composition and lipid metabolism and affect the risk of developing these chronic illnesses. Our group has conducted a randomized clinical trial (LEVA) to evaluate overweight/obese women's ability to make longterm lifestyle changes during the postpartum (pp) period, under ideal study conditions. Physiological mechanisms for weight reduction were investigated with precise methodology. However, effectiveness studies under different conditions are crucial for the development of effective programs for the Primary Health Care sector. Hence, the interest for translational research that brings results from clinical trials to the Primary Health Care sector has increased. The aim of this effectiveness-study is to investigate if dietary restrictions pp lead to significantly greater weight reduction among overweight/obese women, compared to no intervention, in a longterm perspective. In total 106 women will be recruited 10 wk pp and randomized into 1) control group; 2) dietary restrictions in individualized intervention during 12 wks. One and two years pp long term effects are evaluated. Positive results may be integrated into usual practice after the study ends.

ELIGIBILITY:
Inclusion Criteria * BMI at 10 w postpartum >= 27.0

Exclusion Criteria

*Serious disease in mother or child

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2012-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
body weight | 1 and 2 yrs post intervention start

SECONDARY OUTCOMES:
Cost-effectiveness | 1 and 2 years post intervention start

OTHER OUTCOMES:
Reported dietary intake | 1 and 2 yrs post intervention start
  Reported dietary intake by 24 hr recall
Physical activity | 1 yr after start of intervention
  Step counter worn during 5 days
Quality of Life as measured by two validated scales | 1 and 2 yrs after intervention start
  Participants fill in EQ-5D, which is a validated scale often used to calculate QoL
TLC, Transformative Lifestyle Change | At start and end of intervention
  Questions on TLC
Quality of Life as measured by SF-36 | 1 and 2 years after intervention start
  participants fill in SF-36, which is a validated scale, to calculate QoL

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Närhälsan Majorna, Gothenburg
  - Antenatal and child care, Lerum

REFERENCES:
- [Derived] Hagberg L, Winkvist A, Brekke HK, Bertz F, Hellebo Johansson E, Huseinovic E. Cost-effectiveness and quality of life of a diet intervention postpartum: 2-year results from a randomized controlled trial. BMC Public Health. 2019 Jan 8;19(1):38. doi: 10.1186/s12889-018-6356-y. PMID 30621673
- [Derived] Huseinovic E, Bertz F, Leu Agelii M, Hellebo Johansson E, Winkvist A, Brekke HK. Effectiveness of a weight loss intervention in postpartum women: results from a randomized controlled trial in primary health care. Am J Clin Nutr. 2016 Aug;104(2):362-70. doi: 10.3945/ajcn.116.135673. Epub 2016 Jul 13. PMID 27413127